CLINICAL TRIAL: NCT05280522
Title: Influence of Neuromuscular Electrical Stimulation on Pain
Brief Title: Pain Inhibition With Neuromuscular Electrical Stimulation
Status: Completed | Type: Observational
Sponsor: University of New England (Other)
Responsible Party: Sponsor
Other Study IDs: 18.09.05-003
Record Dates: First submitted 2022-02-14; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Healthy Participants
Keywords: Transcutaneous Electric Nerve Stimulation; Noxious Electrical Stimulation; Pain Threshold; Muscle Contraction; Muscle Weakness; Pain Management; Quadriceps; Strength; Pain Inhibition
MeSH Terms: conditions — Muscle Weakness; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Repeated Measures Experiment: Participants are positioned in an isokinetic dynamometer (Biodex System 4 Isokinetic Dynamometer , Biodex Medical Systems, Inc., Shirley, NY) with the knee flexed to approximately 90 degrees. After 3-4 submaximal warm up contractions, participants generate maximum knee extension force while vigorous verbal encouragement is provided. Two trials are collected with 30 seconds between trials. The maximum forces from the 2 trials is used to determine the target force of 20% MVIC used for the volitional and NMES contractions and to normalize the force of the muscle contractions.
  Interventions: Other: Volitional Contractions (VOL); Device: Neuromuscular Electrical Stimulation (NMES); Device: Noxious Electrical Stimulation (NXES)

INTERVENTIONS:
Other: Volitional Contractions (VOL) — Participants are provided visual feedback showing the 20% MVIC force and instructed to produce the target force for 10 s then relax for 50 s. The timing is provided by the research personnel until 10 contractions are completed. Participants rate their pain during each contraction on a visual analog scale. The pain ratings are averaged across all 10 contractions and the average is used in the analysis.
Device: Neuromuscular Electrical Stimulation (NMES) — Participants are instructed to relax throughout the NMES contractions. The amplitude of the stimulation is increased until 20 percent MVIC force is achieved and the amplitude is recorded. The timing of the NMES is 12 s on: 50 s off for 10 contractions. The on-time included a 2s ramp up to the target amplitude. Participants rate their pain during each contraction on a visual analog scale. The pain ratings were averaged across all 10 contractions and the average was used in the analyses.
Device: Noxious Electrical Stimulation (NXES) — The intensity of the electrical stimulation is increased slowly over 30 s to the maximum tolerated level. Trains of NXES are delivered at the maximum tolerated intensity with a timing ratio of 12 s on: 50 s off for a total of 10 trains. The on-time included a 2s ramp up to the target amplitude. Participants rate the pain during each contraction on a visual analog scale. The pain ratings were averaged across all 10 trains of NXES and the average is used in the analyses.

SUMMARY:
The purpose of this study is to demonstrate the pain relieving effect of neuromuscular electrical stimulation that is applied for the purpose of increasing muscle force output.

DETAILED DESCRIPTION:
Electrical stimulation (ES) is used by physical therapists during treatment of many conditions including muscle weakness and pain. Neuromuscular electrical stimulation (NMES) is used to produce strength gains, but it is uncomfortable. The discomfort is thought to limit its acceptability by patients. Transcutaneous electrical stimulation (TENS) is the application of ES for pain relief. The intensity of TENS is strong but comfortable. The nervous system modulates pain in many ways, and one way that it can inhibit pain is through conditioned pain modulation; the "pain inhibits pain" phenomenon. Painful experiences can elicit inhibitory mechanisms that actually reduce pain. This study is designed to demonstrate that NMES elicited muscle contractions produce pain relieving effects that will benefit patients over and above the strengthening effects. Participants will be healthy young (18-30 years of age) who will rate their pain and undergo bilateral quantitative sensory testing of pressure pain over the right quadriceps tendon. They will experience three conditions: volitional contractions at 20 percent of the maximum voluntary isometric contraction (MVIC) force, electrically elicited contractions at 20 percent MVIC, and noxious electrical stimulation (NXES) at maximum tolerated intensity applied to the patella to prevent muscle contraction. Ten contractions or trains of stimulation will be applied at a ratio of 10 seconds on 50 seconds off to replicate the typical application of NMES for muscle strengthening. The order of the conditions will comprise: volitional contractions and NXES will be applied in a random order followed by NMES contractions. NMES was applied last to reduce any influence of muscle fatigue. Pressure pain thresholds (PPT) will be measured before and after each condition in both knees and the middle finder by applying pressure at a rate of 30 kilopascal/s. Participants will indicate immediately when the pressure turns to pain and the pressure will be recorded as their pain threshold. This will be repeated 3 times and the average of the last 2 measurements will be used in the analysis. Participants will rate their pain during the conditions using an 11-point visual analog scales in which 0= no pain and 10= the worst pain imaginable. Testing will take place over two sessions, in the Motion Analysis Laboratory of the University of New England separated by at least one hour. In session 1, participants will be familiarized with any procedures that could cause pain including pressure pain threshold testing, NMES elicited muscle contractions and noxious stimulation. The MVIC force of the quadriceps will also be measured and used to determine the goal force output for the volitional and electrically elicited contractions of 20 percent MVIC. In session 2, participants will undergo the testing procedures, each separated by at least 1 hour.

ELIGIBILITY:
Inclusion Criteria:

Young, healthy men and women between 18-30 years of age

Exclusion Criteria:

* high blood pressure or heart problems;
* Type II diabetes;
* Injury in the last 12 months to your feet, legs, back or spine that required the care of a medical professional;
* pain in the past 6 months that has lasted more than a few days;
* fibromyalgia or other chronic pain condition;
* neurological problems such as stroke;
* dizziness or unexplained falls;
* problems with blood vessels or circulation or skin sensation;
* cancer
* are or could be pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women between 18-30 years of age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Pain Inhibition | day 2
  Pain inhibition will be assessed as the difference in pressure pain threshold (PPT) before and 15 minutes after each condition. PPT will be measured with a pain pressure algometer (Algomed, Medco, Durham, NC). Pressure will be applied over the quadriceps tendon 1 cm proximal to the patella through a 1.0 cm diameter tip at a rate of 30 kilopascals/second. Using a standard script, participants are asked to indicate when the sensation changes from deep pressure to pain. PPTs will be measured at the right (treatment) knee, as well as the contralateral knee and the distal phalanx of the middle finger of the right hand. Three consecutive PPTs will be measured at each site, with ≥ 30 s between each measurement. The last 2 measurements will be averaged and used in the analysis. The change in PPT before and after each condition will comprise the magnitude of pain inhibition.

SECONDARY OUTCOMES:
Pain Ratings | day 2
  Participants will rate their pain during the conditions using a 100 mm visual analog scales in which 0= no pain and 100= the worst pain imaginable. Pain ratings from the 10 contractions or trains of NXES will be averaged and the average will be used in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S Rudolph, PT, PhD, Principal Investigator — University of New England Physical Therapy
Locations (1):
- University of New England Motion Analysis Lab, Portland, Maine, United States